CLINICAL TRIAL: NCT05010486
Title: Prevalence of Sexual Dysfunction After Rectal Surgery and Patient Satisfaction of Preoperative Discussions
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: USherbrooke2
Record Dates: First submitted 2021-08-02; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Sexual Dysfunction; Rectal Surgery; Patient Satisfaction
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: rectal surgery

SUMMARY:
Sexual dysfunction after rectal surgery varies widely in the literature. Prevalence of sexual dysfunction before surgery and desire of patient to treat this condition is also not well established.

Objectives of this prospective cohort study were to determine prevalence of sexual dysfunction with a questionnaire before and after surgery. Patient's satisfaction and quality of life were also collected regarding preoperative information given.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 and 65 years old
* Will undergo one of the following surgeries in the 12 months after the initial visit:

  * Low anterior resection
  * Abdominoperineal resection with end colostomy
  * Total proctocolectomy with ileostomy
  * Total proctocolectomy with ileoanal reservoir
  * Proctectomy
* Having had a sexual intercourse in the 4 weeks prior to the initial visit
* Having the desire to maintain sexual activities in the post-operative period

Exclusion Criteria:

* Tadalafil allergy/hypersensitivity
* Having received treatment for erectile dysfunction or medical treatment in the 4 weeks prior to the initial visit
* Active consumption of nitrate derivatives (NO)
* History of non-arteritic ischemic optic neuropathy
* Severe renal or hepatic insufficiency
* Stroke in the last 6 months
* Myocardial infarction in the last 3 months
* Unstable angina pectoris or angina pectoris during sexual relations
* Cardiac insufficiency Class ≥ 2 in the last 6 months
* Uncontrolled arrhythmia, hypotension or hypertension

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — gender identity
Study Population: Male patients between 18 and 65 years who will have a rectal surgery at the Centre Hospitalier Universitaire de Sherbrooke
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of sexual dysfunction after rectal surgery | 3 years
  Prevalence of sexual dysfunction will be determined with a validated questionnaire on erectile dysfunction (ED). The International Index of Erectile Dysfunction-5 (IIEF-5) focuses on ED; therefore, it only includes the first 5 questions of the IIEF-15. Each item is scored on a 5-point Likert-type ascending scale with a total score between 1 and 25, where a score of 22 and above corresponds to normal erectile function.

SECONDARY OUTCOMES:
Patient satisfaction | 3 years
  Patient satisfaction regarding pre-operative information about the possible side-effects of surgery was assessed with a phone call 1 month after surgery. The quality of the information and the importance given to the possible side-effects of surgery, such as ED, were measured according to the patients' perspective on a 1 to 5 Likert-type ascending scale and a "yes or no" type of response.
Sexual dysfunction and quality of life | 3 years
  Quality of life was measured by the Quality of Life Enjoyment and Satisfaction (LES) Questionnaire Short Form (Q-LES-Q-SF), a 16-item derivative from the Q-LES-Q, a 93-item questionnaire. Patients' satisfaction was evaluated by a 5-point Likert-type ascending scale. The first 14 questions were scored from 14 to 70 points in total, while the last two items addressing medication and overall quality of life were represented by two independent scores of 5 points. Q-LES-Q-SF scores were measured at baseline during the first clinical visit as well as 1 month, 6 months, and 12 months after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie McFadden, M.D, Principal Investigator — Université de Sherbrooke